CLINICAL TRIAL: NCT00221247
Title: Acupuncture as Complementary Therapy for Cerebral Palsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Burris Duncan, Professor of Pediatrics & Public Health, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC #04-126; ADCRC: No. 9-039 (Other Grant/Funding Number: ADCRC); Commission contract No.9001 (Other: Commission)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; acupuncture
MeSH Terms: conditions — Cerebral Palsy | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Intensely administered (5 times per week for 12wk) physical therapy, occupational therapy, and hydrotherapy with acupuncture
  Interventions: Procedure: Acupuncture
- Group 2 (No Intervention): Intensely administered (5 times per week for 12wk) physical therapy, occupational therapy, and hydrotherapy without acupuncture

INTERVENTIONS:
Procedure: Acupuncture — acupuncture
  Arms: Group 1

SUMMARY:
Background: Cerebral palsy (CP) is the most frequent cause of childhood disability in the US. Nevertheless, current standard of care for CP in the U.S. is to a large extent ineffective. The Chinese, on the other hand, claim to have an exceptionally high response rate with the administration of an integrated package of care that includes the combination of intense 'conventional' therapies and acupuncture. Despite numerous anecdotal reports, this claim has not yet been tested in a rigorous scientific way. Objective: To determine the effectiveness of acupuncture when used as an adjunct to intense 'conventional' physical, occupational, and hydro- therapies to improve function and quality of life in children with spastic CP. Hypotheses: (1) Adjunctive acupuncture therapy will improve the gross and fine motor function and the health related quality of life of children with spastic CP more than intense 'conventional' therapies alone. (2) The level of persistence of gross and fine motor function and health related quality of life achieved with adjunctive acupuncture administered in combination with intense 'conventional' therapies will be higher than those achieved with intense 'conventional' therapies alone. Design: A parallel, two-arm, prospective, evaluation-blind, pragmatic, non-inferiority, randomized controlled clinical trial (RCT). Setting: This international collaborative study will be conducted at two different localities: (1) At the Beijing Children's Hospital (BCH), where participants' recruitment, intervention therapies, videotape evaluation, and data collection will be done, and (2) At the University of Arizona, where scoring of the videotape evaluations and data analyses will be done, and from where logistic support will be provided to assure the scientific integrity of the study. Population: Approximately 100 children between the ages 1 and 6 years with spastic CP. Intervention: Concurrent administration of acupuncture with intense 'conventional' therapies at the outset of the study vs. sequential administration of both components. Outcomes: 'Gross Motor Function', 'Fine Motor Function', 'Range of Motion', 'Level of Motor Involvement', and 'Health-Related Quality of Life' measured at times 0,4,8,12,24,and 36 weeks. Evaluation: Independent blinded evaluation with respect to the type of the intervention and the stage of the therapeutic schedule done in the U.S. based on videotapes filmed in China. Data management: Web-based data center and intersite-networking infrastructure. Data analyses: Intention to treat analysis supplemented by linear mixed effects models with nested grouping factors. Significance and future directions: If the hypotheses are confirmed the study would lay the groundwork for future research, and impact clinical practice and health care policy as related to CP therapy.

DETAILED DESCRIPTION:
The proposed study is a parallel, two-arm, prospective, evaluation-blind, randomized controlled clinical trial (RCT). It has been designed to examine the effectiveness of acupuncture when used as an adjunct to intense 'conventional' physical, occupational, and hydro- therapies to improve function and quality of life in children with spastic cerebral palsy (CP). This international collaborative study will be conducted at two locations: (1) At the Beijing Children's Hospital (BCH), where participants' recruitment, intervention therapies, videotape evaluation, and data collection will be done, and (2) At the University of Arizona, where scoring of the videotape evaluations and data analyses will be done, and from where logistic support will be provided to assure the scientific integrity of the study. The specific aims of the proposed study are:

Specific Aim #1: To compare the outcomes achieved after 12 weeks of acupuncture administered concurrently with intense 'conventional' therapies (physical, occupational, and hydro-therapies) to those achieved with intense 'conventional' therapies alone in the management of children with spastic CP.

Hypothesis #1: Adjunctive acupuncture administered concurrently with intense 'conventional' therapies will improve the gross and fine motor function and the health related quality of life of children with spastic CP more than intense 'conventional' therapies alone, as determined by standardized measures (see pgs. 20-22).

Specific Aim #2: To examine the short and intermediate term persistence of any changes in the outcomes achieved with acupuncture administered concurrently with intense 'conventional' therapies (physical, occupational, and hydro-therapies) to those achieved with intense 'conventional' therapies alone in the management of children with spastic CP.

Hypothesis #2: When compared three months after termination of therapy, the level of gross and fine motor function and health related quality of life achieved with acupuncture administered concurrently with intense 'conventional' therapies (physical, occupational, and hydro-therapies) will be higher than those achieved with intense 'conventional' therapies alone.

Taking advantage of the fact that ethically all the Chinese children with spastic CP who would participate in this study ought to receive acupuncture at one point or another as part of their care (see pg. 12) we propose, as a secondary aim, to begin to examine whether the timing of the administration of adjunctive acupuncture in relation to the timing of the administration of intense 'conventional' therapies has any effect on the outcomes, as determined by standardized measures.

It is to be emphasized, that this study does not aim primarily at testing sequence effects related to the most appropriate timing of administration of adjunctive acupuncture in the treatment of children with spastic CP since a) it must first be examined whether acupuncture has any effect at all in this population, and b) testing sequence effects would greatly complicate the design of such a study to a point where it may render it not feasible. Rather, we are simply taking advantage of the ethical obligation to provide every participant with acupuncture at some point in time (not because it is proven from an efficacy standpoint but because it is the standard of care in China) so as to begin to explore any potential temporal relationships between administration of adjunctive acupuncture and outcomes. For example, since Group 1 would receive adjunctive acupuncture concurrently with intense 'conventional' therapies whereas Group 2 would receive adjunctive acupuncture therapy subsequently to intense 'conventional' therapies (see Figure 1 on pg. 11), the design allows to begin to explore whether adjunctive acupuncture administered subsequent to intense 'conventional' therapies may have a booster effect on the degree of gross and fine motor function and health related quality of life of children with spastic CP.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 12 and 72 months.
* Children with a diagnosis of spastic cerebral palsy (CP) or mixed type CP where spasticity is the dominant feature.

Exclusion Criteria:

* Age - Any child with CP who is younger than 12 months or older than 72 months.
* Etiology - Any damage to the CNS that either (a) is not static in nature, such as degenerative or progressive central nervous disorders, or (b) occurred after the first year of life, or (c) any child who has a phenotypic pattern suggesting a chromosomal abnormality (e.g., trisomy 13 or 18).
* Diagnosis - Children for whom the diagnosis of spastic CP or mixed-type CP with spasticity as the dominant feature cannot be established with absolute certainty, or children with dyskinetic CP. Rationale - To assure subject homogeneity, in cases in which there is disagreement between the physicians with respect to the diagnosis of a child, even if one of the physicians feels certain that a child has spastic CP, the children would be automatically excluded.
* Co-morbidities - Medical conditions, whether acute or chronic, for which acupuncture or intense 'conventional' therapies are considered contraindicated. Rationale - assuring participants' safety.
* Co-interventions - Any child receiving or scheduled to receive treatment(s) during the study period that may confound the results (e.g., an orthopedic or neurosurgical procedure, Botulinum toxin injections, a Baclofen pump or hyperbaric oxygen treatment). Rationale -To avoid a threat to causal inferences.
* Parallel participation in another CP clinical trial. Rationale - To avoid pragmatic and ethical issues that may arise as a result of a conflict of interests and limited resources.

Ages: 12 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2004-10; Primary Completion 2008-03 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burris Duncan, M.D., Principal Investigator — The University of Arizona, Department of Pediatrics
Locations (2):
- The University of Arizona, Department of Pediatrics, Tucson, Arizona, United States
- Beijing Children's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Duncan B, Shen K, Zou LP, Han TL, Lu ZL, Zheng H, Walsh M, Venker C, Su Y, Schnyer R, Caspi O. Evaluating intense rehabilitative therapies with and without acupuncture for children with cerebral palsy: a randomized controlled trial. Arch Phys Med Rehabil. 2012 May;93(5):808-15. doi: 10.1016/j.apmr.2011.12.009. PMID 22541308
- [Derived] Wu Y, Zou LP, Han TL, Zheng H, Caspi O, Wong V, Su Y, Shen KL. Randomized controlled trial of traditional Chinese medicine (acupuncture and tuina) in cerebral palsy: part 1--any increase in seizure in integrated acupuncture and rehabilitation group versus rehabilitation group? J Altern Complement Med. 2008 Oct;14(8):1005-9. doi: 10.1089/acm.2007.0756. PMID 18990048